CLINICAL TRIAL: NCT07341724
Title: Telemedicine for Evaluating Dry Eye Disease (DED) Using a Mobile Phone-Attached Portable Automatic Ocular Surface Imaging Device (PAOSID): A Patient-Operated Diagnostic and Continuous Ocular Surface Monitoring (COSM) System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2025-0263; 2025-0263 (Other: SingHealth CIRB)
Record Dates: First submitted 2025-12-21; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye; Dry Eye Disease (DED)
Keywords: PAOSID; Dr EYE
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient diagnose with Dry Eye Disease (Other)
  Interventions: Diagnostic Test: Dr Eye
- Healthy subject (Other)
  Interventions: Diagnostic Test: Dr Eye

INTERVENTIONS:
Diagnostic Test: Dr Eye — Portable automatic ocular surface imaging device (PAOSID) that attaches to a mobile phone has been developed. This device uses three types of light including white, infrared, and cobalt blue light to capture clear images and videos of the eye's surface.
  It also has a smart system that automatically takes high-quality images, allowing patients to use it at home independently. This device may help detect early signs of DED and monitor eye health more easily.

SUMMARY:
Dry eye disease (DED) is a common eye condition that is becoming more widespread. Detecting it early, keeping track of its progression, and following up regularly can help protect vision and prevent serious complications. However, due to a shortage of ophthalmologists, limited access to eye care services, and disparities in care quality, many patients receive infrequent or insufficient clinical consultations.

To address these needs, a portable automatic ocular surface imaging device (PAOSID) that attaches to a mobile phone has been developed. This device uses three types of light including white, infrared, and cobalt blue light to capture clear images and videos of the eye's surface.

It also has a smart system that automatically takes high-quality images, allowing patients to use it at home independently. This device may help detect early signs of DED and monitor eye health more easily.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed as DED by experienced ophthalmologists, based on the TFOS DEWS II (The Tear Film and Ocular Surface Society Dry Eye Workshop II) guidelines,(19) as well as healthy individuals with no ocular conditions who voluntarily agreed to participate in the study;
2. Participants, or their companions or caregivers, who are willing and able to use the study smartphone to capture relevant eye images and videos;
3. Aged 21 years or older;
4. Provide informed consent.

Exclusion Criteria:

1. Participants with ocular surface disorders other than DED that may affect the appearance of the ocular surface (e.g., pterygium, keratitis, corneal scarring) or with any organic pathologies impacting vision (e.g., cataracts, glaucoma, retinal diseases).
2. Patients currently wearing scleral lenses or bandage contact lenses.
3. Significant changes in the ocular images since diagnosis due to factors such as postdiagnostic treatment;
4. Unable to cooperate with the PAOSID, such as due to a serious mental illness or brain damage causing loss of limb control;
5. Eyes with previous or active corneal diseases such as infectious keratitis, corneal opacity or dystrophy;
6. Eyes with active inflammation or infection.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to study the diagnostic accuracy of remote Dry Eye Disease (DED) diagnosis using a portable automatic ocular surface imaging device (PAOSID), as compared with standard clinical DED diagnosis. | From enrollment to end of visit 1, estimated 1 hour (One Time Visit)

SECONDARY OUTCOMES:
The secondary objectives: diagnostic consistency of remote Dry Eye Disease (DED) diagnosis using a portable automatic ocular surface imaging device (PAOSID), as compared with standard clinical DED diagnosis. | From enrollment to end of visit 1, estimated 1 hour (One Time Visit)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore Eye Research Institute